CLINICAL TRIAL: NCT02626858
Title: Optimizing the Delineation of the Tumour Bed in Breast Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s54017
Record Dates: First submitted 2015-09-28; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- extra treatment planning CT-scan (Other): Extra pre-operative CT-scan for treatment planning in RT
  Interventions: Device: extra treatment planning CT-scan

INTERVENTIONS:
Device: extra treatment planning CT-scan — Beside the standard post-operative CT-scan, an extra pre-operative CT-scan is performed.

SUMMARY:
The aim of the present study is:

1. to verify whether the delineation of the tumour bed, based on the combination of the visible postoperative changes and the position of the surgical clips on a CT scan in treatment position acquired 1 week before the start of the radiotherapy (RT), provides an accurate localisation of the boost volume compared to the localisation of the tumour on a pre-operative CT-scan.
2. to document the changes that occur in the tumour bed as seen on a CT scan as a function of the delay between surgery and radiotherapy.
3. to determine the ideal number and the positioning of the clips needed to reproduce the best treatment volume for the boost.
4. to propose new guidelines for tumour bed definition and delineation based on the study findings.

DETAILED DESCRIPTION:
Start of the study: february 2012

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer patients, without metastases, who will undergo breast conserving surgery and probably will receive adjuvant chemotherapy and thereafter radiotherapy.

Exclusion Criteria:

* Metastases at time of diagnosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the interobserver variability (IOV) (%) of the delineated Clinical Target Volume (CTV) boost (cm3) with and without the fusion of the pre-operative CT-scan. | 2 years
the volume of the delineated CTVboost (cm3) with and without the fusion of the pre-operative CT-scan. | 2 years

SECONDARY OUTCOMES:
the correlation of the Cavity Visibility Scale (CVS) to volume changes and IOV | 2 Years
the volume changes over time (in case of adjuvant chemotherapy) | 2 years
the usefulness of the surgical clips assessed by the 6 observers. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Weltens, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium